CLINICAL TRIAL: NCT00244452
Title: A Multinational, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Investigate the Efficacy, Safety and Duration of Effect of a Single Administration of Various Doses of Cetrorelix SR in Subjects With Histologically Confirmed Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Gereon Raddatz, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S184.2.101; 2004-004739-67
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Endometriosis
Keywords: Endometriosis; Cetrorelix; Hormone; Symptoms relief; Safety; Tolerability; Pharmacodynamic; Pharmacokinetic
MeSH Terms: conditions — Endometriosis | interventions — cetrorelix

INTERVENTIONS:
Drug: Cetrorelix

SUMMARY:
Identify effective doses of cetrorelix SR in the treatment of symptoms of endometriosis, describe dose effect relationship and duration of symptom relief

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female,
* history of regular menstrual periods,
* any of the symptoms dysmenorrhea,
* dyspareunia or pelvic pain assessed as moderate to severe,
* endometriosis confirmed by histology within 36 months,
* use of barrier contraception throughout the study

Exclusion Criteria:

* Insufficient wash out period for other endometriosis treatments,
* resection or destruction of endometriotic lesions less than 12 weeks prior to screening,
* need for strong opioid analgesics,
* need for immediate surgical treatment of endometriosis,
* any condition that interferes with adherence to study procedures or study assessments

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (57):
- Australia (4):
  - Site 6101, Clayton
  - Site 6103, Nedlands
  - Site 6104, Randwick
  - Site 6102, Sydney
- Belgium (3):
  - Site 3201, Aalter
  - Site 3202, Brussels
  - Site 3203, Leuven
- Bulgaria (6):
  - Site 3501, Sofia
  - Site 3502, Sofia
  - Site 3503, Sofia
  - Site 3504, Sofia
  - Site 3505, Sofia
  - Site 3506, Sofia
- Germany (5):
  - Site 4904, Berlin
  - Site 4905, Dresden
  - Site 4903, Heidelberg
  - Site 4901, Herne
  - Site 4902, Tübingen
- Romania (10):
  - Site 4000, Bucharest
  - Site 4001, Bucharest
  - Site 4002, Bucharest
  - Site 4004, Bucharest
  - Site 4005, Bucharest
  - Site 4006, Bucharest
  - Site 4007, Bucharest
  - Site 4009, Bucharest
  - Site 4008, Constanța
  - Site 4003, Craiova
- Russia (16):
  - Site 0701, Moscow
  - Site 0901, Moscow
  - Site 0902, Moscow
  - Site 0903, Moscow
  - Site 0904, Moscow
  - Site 0905, Moscow
  - Site 0906, Moscow
  - Site 0907, Moscow
  - Site 0908, Moscow
  - Site 0909, Moscow
  - Site 0702, Saint Petersburg
  - Site 0703, Saint Petersburg
  - Site 0704, Saint Petersburg
  - Site 0705, Saint Petersburg
  - Site 0706, Saint Petersburg
  - Site 0707, Saint Petersburg
- South Africa (5):
  - Site 2705, Bloemfontein
  - Site 2703, Cape Town
  - Site 2702, Centurion
  - Site 2701, Roodepoort
  - Site 2704, Roodepoort
- Ukraine (8):
  - Site 3805, Dnipro
  - Site 3801, Donetsk
  - Site 3803, Kiev
  - Site 3806, Kiev
  - Site 3807, Kiev
  - Site 3808, Kiev
  - Site 3802, Odesa
  - Site 3804, Zaporizhzhya